CLINICAL TRIAL: NCT00518791
Title: Integrated Multidisciplinary Care for Parkinson's Disease: a Controlled Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting Nuts Ohra (Other); Porticus (Unknown)
Responsible Party: Dr M Munneke, UMC St Radboud, Neurology
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2010-IP5.1
Record Dates: First submitted 2007-08-20; First posted 2007-08-21 (Estimated); Last update posted 2010-11-05 (Estimated); Status verified 2010-10

CONDITIONS: Parkinson's Disease
Keywords: Integrated health care system; Treatment effectiveness; Cost effectiveness; Program evaluation
MeSH Terms: conditions — Parkinson Disease | interventions — Patient Care Team

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- I (Experimental): Multidisciplinary Care
  Interventions: Other: Multidisciplinary Care
- II (Other): Usual Care
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Multidisciplinary Care — A comprehensive individualised assessment by a dedicated multidisciplinary team (Multidisciplinary Assessment Center) and subsequent treatment by specifically trained health professionals (ParkinsonNet).
  Arms: I
Other: Usual Care — No altered organisation of care
  Arms: II

SUMMARY:
The aim of the present study is to evaluate the (cost) effectiveness of a new health care system in which an individualised multidisciplinary assessment is given to patients with Parkinson's Disease(PD)in combination with treatment by a dedicated team of specifically trained health professionals, compared to usual care. Overall, we anticipate to gain more insight in the clinical effectiveness and health care costs of multidisciplinary treatment in PD.

DETAILED DESCRIPTION:
PD is a complex disorder, with motor as well as non-motor symptoms. Despite the complexity of PD, management of the disease is often 'monodisciplinary' since most patients are only treated by a neurologist. Stimulating compensatory strategies by allied health professionals might offer additional therapeutic relief, but this assumption is mainly based on theoretical arguments and expert opinion. Even less is known about the claim that a multidisciplinary team of multiple professionals active in complementary domains (e.g. physiotherapy, occupational therapy and speech therapy) is superior to management by each of these professionals alone.

This study anticipates to provide more insight in the clinical effectiveness and health care costs of multidisciplinary treatment in PD. Therefore, our multidisciplinary care concept (a comprehensive assessment by a dedicated multidisciplinary team and subsequent treatment by specifically trained health professionals) that is tailored to the patients' individual needs will be compared to usual care in terms of effectiveness and costs.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Idiopathic PD, diagnosed according to the Brain Bank Criteria of the UK Parkinson's Disease Society
* Regular control by the neurologist
* Living independently in the community
* Able to complete the trial questionnaires

Exclusion Criteria:

* Atypical parkinsonian syndromes
* Hoehn and Yahr stage 5
* Severe cognitive impairment (MMSE<24)
* Presence of other neurological disorders
* Severe co-morbidity (e.g. cancer)
* Planned surgical procedure for PD within the intervention period
* Patients who have already visited the Multidisciplinary Assessment Center

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 301 (Actual)
Dates: Start 2007-08; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
Parkinson's Disease Quality of Life Questionnaire (PDQL) | 8 months
AMC Linear Disability Score (ALDS) | 8 months

SECONDARY OUTCOMES:
SF-36 (secundary;utility score) | 8 months
UPDRS Motor Examination (part III)(secondary) | 4 months
UPDRS Complications of therapy (part IV)(tertiary) | 4 months
SPDDS(tertiary) | 8 months
Modified MACTAR scale(tertiary) | 8 months
Parkinson Activity Scale(tertiary) | 4 months
Costs (secondary) | 8 months
Frequency of falls (tertiary) | 8 months
Freezing of Gait Questionnaire (tertiary) | 8 months
Falls Efficacy Scale (tertiary) | 8 months
Non-Motor Symptom Assessment Scale and Quest for Parkinson's Disease (tertiary) | 8 months (Quest) and 4 months (Scale)
Hospital Anxiety and Depression Scale (tertiary) | 8 months
Caregiver burden assessed with BELA-A-k (secondary), SF-36 (tertiary), and HADS (tertiary) | 8 months

CONTACTS AND LOCATIONS:
Overall Officials: Marten Munneke, PhD, Principal Investigator — UMC St Radboud; Bastiaan R Bloem, MD, PhD, Principal Investigator — UMC St Radboud; Marjolein A van der Marck, MSc, Principal Investigator — UMC St Radboud
Locations (6):
- Netherlands (6):
  - Ziekenhuis Groep Twente, Twenteborg Ziekenhuis, Almelo
  - Ziekenhuis Rijnstate, Arnhem
  - Wilhelmina Ziekenhuis Assen, Assen
  - Ziekenhuis Groep Twente, Streekziekenhuis Midden-Twente, Hengelo
  - Medisch Centrum Leeuwarden, Leeuwarden
  - Canisius Wilhelmina Ziekenhuis, Nijmegen

REFERENCES:
- [Derived] van der Marck MA, Munneke M, Mulleners W, Hoogerwaard EM, Borm GF, Overeem S, Bloem BR; IMPACT study group. Integrated multidisciplinary care in Parkinson's disease: a non-randomised, controlled trial (IMPACT). Lancet Neurol. 2013 Oct;12(10):947-56. doi: 10.1016/S1474-4422(13)70196-0. Epub 2013 Aug 27. PMID 23988337